CLINICAL TRIAL: NCT01367392
Title: Confirmation of Clinical Effectiveness and Safety of CT-guided Needle Placement in the Liver With the Aid of the ActiSight Needle Guidance System
Brief Title: Effectiveness and Safety of CT-guided Needle Placement in the Liver With the Aid of the ActiSight Needle Guidance System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ActiViews Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ACST-2011-1
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Accurate Navigation to the Lesion
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- interventional procedure (Experimental): The patients undergo the required interventional procedure, biopsy or ablation
  Interventions: Device: biopsy or ablation

INTERVENTIONS:
Device: biopsy or ablation — biopsy or ablation performed as in standard of care with assistance of ActiSight Needle Guidance system

SUMMARY:
The purpose of this study is to confirm the safety and effectiveness of the ActiSight™ Needle Guidance System with CT-guided percutaneous (through the skin) liver biopsies and ablations . The device used in this study is designed to assist the physician in guiding the needle towards the suspected area. This device does not change the procedure of liver biopsy or ablation. The only difference is that a small adhesive pad is placed on the skin and a miniature video camera is attached to the end of the needle. This camera does not enter the body.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female subjects, between the ages of 18 and 80 at the time of enrollment.
* Subjects scheduled for clinically indicated CT guided percutaneous needle placements in the liver who meet the desired target population described above.
* Written informed consent to participate in the study.
* Ability to comply with the requirements of the study procedures.
* Verified home address and phone number to facilitate study follow-up.

Exclusion Criteria:

* Significant coagulopathy that cannot be adequately corrected.
* Subjects who participated in an active stage of any drug, intervention or treatment trial within 30 days of enrollment.
* Subjects with preexisting conditions, which, in the opinion of the investigator, interfere with the conduct of the study.
* Subjects who are uncooperative or cannot follow instructions.
* Mental state that may preclude completion of the study procedure.
* Pregnant or nursing female subjects.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
accuracy | during the procedure
  Frequency of placing the needle at a location suitable for the planned intervention, as determined by the investigator reviewing the CT images.

SECONDARY OUTCOMES:
time | during the procedure
  Total CT-Guided procedure time, starting with scan for entry point planning;
time | during the procedure
  Time required to guide the needle to the target
radiation | during the procedure
  Subject radiation exposure during the procedure
total number of scans | during the procedure
  Number of CT scans during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada